CLINICAL TRIAL: NCT00457054
Title: Functional Connectivity in Mood Regulating Circuit In Bipolar Depression and Mania Before and After Lithium Treatment: An Brain fMRI Study
Brief Title: Functional Connectivity in Mood Regulating Circuit In Bipolar Depression and Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Amit Anand, M.D., Indiana University School of Medicine Department of Psychiatry
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0303-28; 61-869-18
Record Dates: First submitted 2005-09-14; First posted 2007-04-05 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Bipolar Depression
Keywords: Mood Regulating Circuit; Lithium; fMRI
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lithium — starting dose 600 mg increase as tolerated

SUMMARY:
The purpose of this study is to find out what parts of the brain have increased or decreased activity with individuals who have bipolar disorder and how medicine changes this activity in bipolar subjects. Another purpose of this study is to compare data obtained from bipolar depressed subjects with data obtained from healthy subjects. In this study we will measure activity in different parts of the brain, while participants see pictures, using Magnetic Resonance Imaging (MRI) scan. We will do two MRI scans with each subject before and after treatment for eight weeks with a standard bipolar disorder medication called lithium.

DETAILED DESCRIPTION:
Aim 1: Our first aim is to use a novel fMRI experimental paradigm to investigate the pathophysiology of bipolar disorder (BD) in terms of the strength of connectivity (as measured by LFBF correlations) between the different emotion regulating areas of the brain rather than in terms of increase or decrease in localized brain activity.

Specific Aim 2: Our second aim is to investigate whether lithium works by altering the connectivity of areas of the brain implicated in the pathophysiology of BD, thereby leading to changes in the abnormal positive or negative emotional reactions to the environment seen in mania and depression respectively.

Specific Aim 3: Out third aim is to investigate whether patients with the s/s or s/L alleles of the 5-HTTLPR polymorphism will have greater amygdalar activation and decreased cortico-amygdala connectivity compared to patients with L/L genotype. We will also investigate whether lithium treatment differentially affects these fMRI measures in the s/s or s/L and L/L genotypes.

Methods:

We will study unmedicated subjects satisfying DSM-IV criteria for Bipolar Disorder current episode depressed or hypomanic/manic or who are euthymic. Subjects will undergo fMRI before and after 8 weeks of treatment with lithium a mood stabilizer that is known to be effective in both phases of BD. Healthy subjects will have a scan at baseline and after 8 weeks but will not be treated with any medication. We will also test for the serotonin transporter gene (the gene that controls the availability of a chemical called serotonin in the brain), which has been shown to effect how lithium works.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Bipolar Subjects

* Ages 18-60 years and able to give voluntary informed consent.
* Satisfy criteria for Bipolar Depression using the Structured Clinical Interview for Diagnostic and Statistical Manual -4th edition (DSM-IV) (SCID-IV).
* Bipolar depressed subjects: 25-item Hamilton Depression Rating Scale (HDRS) score > 18.Young Mania Rating Score (YMRS)<10.
* Bipolar hypomanic/manic subjects will have a YMRS score>12 and a 25-item HDRS score<10.
* Bipolar Euthymic subjects will have YMRS score < 10 and HDRS score < 10 and would have been euthymic for > 14 days.
* Subjects will be drug and medication free and would have no significant history of medical or neurological illness.
* Satisfy criteria to undergo an MRI scan based on MRI screening questionnaire
* Able to be managed as outpatients for initial assessment and during treatment as ascertained by the following:

  * Symptoms not worsening by more than 10 points on either the HDRS or the YMRS during the course of the study.
  * No danger to self or others.
  * No psychotic symptoms.

Inclusion criteria for Healthy Subjects:

* Ages 18-60 years and able to give voluntary informed consent.
* No history of psychiatric illness or substance abuse or dependence as assessed by SCID for non-patients (SCID-NP).
* No significant family history of psychiatric or neurological illness.
* Not currently taking any prescription or centrally acting medications.
* No serious medical or neurological illness as assessed by history, physical examination and laboratory examination including CBC and blood chemistry.

Exclusion Criteria:

Exclusion criteria for Bipolar Subjects

* Meeting DSM-IV criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, atypical psychosis, mental retardation, or organic mental (including organic mood) disorder.
* Use of neuroleptic past 2 weeks
* Use of antidepressants in the past 2 weeks. If on fluoxetine in the past then should not have been on this medication for 4 weeks.
* Use of mood stabilizers in the past 2 weeks
* Use of benzodiazepines in the past 2 weeks.
* Acutely suicidal or homicidal or requiring inpatient treatment.
* Meeting DSM-IV criteria for other substance dependence within the past year, except caffeine or nicotine. The criteria will be evaluated by interview and urinary toxicology screening initially and on test days.
* Use of alcohol in the past 1 week.
* No serious medical or neurological illness as assessed by physical examination and laboratory examination including complete blood count (CBC) and blood chemistry.
* Current pregnancy or breast feeding.
* Metallic implants.
* Previously known positive Human Immunodeficiency Virus (HIV) blood test as reported by the subject.

Exclusion criteria for Healthy Subjects:

* Under 18 years of age.
* Pregnant or breast feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Comparative activation of amygdala and cortico-amydalar connectivity as measured by fMRI taken at baseline and eight weeks from baseline | 07-03 to 3-07
Improvement of scores on Hamilton Depression Rating Scale given weekly for eight weeks | 07-03 to 3-07

SECONDARY OUTCOMES:
Improvement as measured by the Clinical Global Impression Severity and Improvement Scales given weekly for eight weeks | 07-03 to 3-07
Improvement as measured by the Brief Psychiatric Rating Scale given weekly for eight weeks | 07-03 to 3-07

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Adult Psychiatry Clinic, Indianapolis, Indiana, United States